CLINICAL TRIAL: NCT01464333
Title: Humira® for Subcutaneous Injection Protocol for Special Investigation (Long-term Treatment for Crohn's Disease Patients)
Brief Title: Special Investigation (Long-term Investigation) in Patients With Crohn's Disease
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-170
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Humira: Participants who were prescribed Humira per approved prescribing information of Humira in Japan.

SUMMARY:
This study of Humira will be conducted to obtain information on the safety (especially profile of malignant tumors and serious infections) and effectiveness in patients with Crohn's disease who are receiving Humira for a long period of time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease indicated for Humira treatment with the recommended dosage regimen
* Patients with no past- or present malignant tumors
* Patients who are not currently receiving Humira

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those who are receiving Humira in accordance with its indications for treatment and dosage regimens.
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2011-12-16 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 511 patients enrolled, case report forms were not collected from 7 patients (N = 504). The safety analysis set excluded 115 enrolled patients due to "safety assessment impossible" (N = 389). The efficacy analysis set excluded 79 patients that were included in the safety analysis set due to "efficacy assessment impossible" (N = 310).
Period: Overall Study
Arm/Group | Humira
Started | 389
Completed | 226
Not Completed | 163
Not completed — Adverse Event | 34
Not completed — Lack of Efficacy | 72
Not completed — Withdrawal by Subject | 11
Not completed — Other | 4
Not completed — No Hospital Visit | 42

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Arm/Group | Humira
Number analyzed (Participants) | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 283
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 389

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event was any untoward or unintended symptoms (including abnormal laboratory findings), condition or illness, which are not always related to Humira. Please see Adverse Event section below for more details.
Time Frame: From first dose of Humira up to 3 years
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 389
participants
  Serious Adverse Events | 58
  Non-serious Adverse Events | 104

2. Secondary Outcome: Change in Crohn's Disease Activity Index (CDAI) Score Over Time
Description: The Change in Crohn's Disease Activity Index (CDAI) is used to evaluate the activity of Crohn's disease. The CDAI is calculated on the basis of a one-week evaluation of 8 items and ranges from 0 to about 600. The 8 items are frequency of liquid or very soft stool, abdominal pain, complications of Crohn's disease (e.g., uveitis, arthritis, fistula, and abscess), abdominal mass, hematocrit, body weight, use of antidiarrheals, and general condition. Low scores indicate low activity of Crohn's disease. In general, CDAI scores below 150 represent remission and scores over 450 represent very severe Crohn's disease. A negative change from Baseline indicates improvement.
Time Frame: From first dose of Humira up to 3 years
Population: Efficacy Analysis Set: patients who have assessments at the first administration and the subsequent assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 310
units on a scale
  At first administration: number analyzed (Participants) | 259
  At first administration | 193.68 (103.00)
  Week 4 of administration: number analyzed (Participants) | 226
  Week 4 of administration | 115.17 (72.21)
  Month 3 of administration: number analyzed (Participants) | 185
  Month 3 of administration | 108.43 (80.45)
  Month 6 of administration: number analyzed (Participants) | 161
  Month 6 of administration | 100.29 (84.14)
  Year 1 of administration: number analyzed (Participants) | 162
  Year 1 of administration | 108.81 (83.40)
  Year 1 and Month 6 of administration: number analyzed (Participants) | 146
  Year 1 and Month 6 of administration | 90.86 (71.84)
  Year 2 of administration: number analyzed (Participants) | 123
  Year 2 of administration | 93.90 (75.99)
  Year 2 and Month 6 of administration: number analyzed (Participants) | 113
  Year 2 and Month 6 of administration | 88.92 (76.62)
  Year 3 of administration: number analyzed (Participants) | 96
  Year 3 of administration | 94.89 (81.61)

3. Secondary Outcome: Change In Work Productivity and Activity Impairment (WPAI): Crohn's Disease (CD) Absenteeism Over Time
Description: WPAI: CD is a questionnaire used to evaluate lost productivity due to CD; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Absenteeism (percentage of work time missed due to CD) is calculated as the number of hours of work missed due to CD / (number of hours of work missed due to CD + number of hours worked) * 100. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: From first dose of Humira up to 3 years
Population: Efficacy Analysis Set: patients who have assessments at the first administration and the subsequent assessment
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Humira
Number analyzed (Participants) | 310
percentage of work time missed
  At first administration: number analyzed (Participants) | 118
  At first administration | 30.71 (42.35)
  Week 4 of administration: number analyzed (Participants) | 102
  Week 4 of administration | 11.86 (28.81)
  Month 3 of administration: number analyzed (Participants) | 84
  Month 3 of administration | 11.12 (28.17)
  Month 6 of administration: number analyzed (Participants) | 72
  Month 6 of administration | 7.04 (22.35)
  Year 1 of administration: number analyzed (Participants) | 63
  Year 1 of administration | 8.34 (24.94)
  Year 1 and Month 6 of administration: number analyzed (Participants) | 41
  Year 1 and Month 6 of administration | 10.34 (28.03)
  Year 2 of administration: number analyzed (Participants) | 30
  Year 2 of administration | 5.49 (19.54)
  Year 2 and Month 6 of administration: number analyzed (Participants) | 29
  Year 2 and Month 6 of administration | 7.33 (23.26)
  Year 3 of administration: number analyzed (Participants) | 22
  Year 3 of administration | 4.69 (21.30)

4. Secondary Outcome: Change in WPAI: CD Presenteeism Over Time
Description: WPAI: CD is a questionnaire used to evaluate lost productivity due to CD; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Presenteeism (percentage of impairment while working due to CD ) is calculated as the patient's rating of how much CD affected productivity while working (0 = no effect; 10 = completely prevented from working) / 10 * 100. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: From first dose of Humira up to 3 years
Population: Efficacy Analysis Set: patients who have assessments at the first administration and the subsequent assessment
Measure: Mean (Standard Deviation); unit: Percent impairment while working
Arm/Group | Humira
Number analyzed (Participants) | 310
Percent impairment while working
  At first administration: number analyzed (Participants) | 112
  At first administration | 38.13 (32.87)
  Week 4 of administration: number analyzed (Participants) | 92
  Week 4 of administration | 24.57 (27.07)
  Month 3 of administration: number analyzed (Participants) | 77
  Month 3 of administration | 24.03 (26.91)
  Month 6 of administration: number analyzed (Participants) | 65
  Month 6 of administration | 19.85 (27.47)
  Year 1 of administration: number analyzed (Participants) | 63
  Year 1 of administration | 22.22 (28.93)
  Year 1 and Month 6 of administration: number analyzed (Participants) | 39
  Year 1 and Month 6 of administration | 27.69 (32.80)
  Year 2 of administration: number analyzed (Participants) | 27
  Year 2 of administration | 21.85 (24.18)
  Year 2 and Month 6 of administration: number analyzed (Participants) | 25
  Year 2 and Month 6 of administration | 20.40 (29.08)
  Year 3 of administration: number analyzed (Participants) | 19
  Year 3 of administration | 14.21 (24.11)

5. Secondary Outcome: Change in WPAI: CD Overall Work Impairment Over Time
Description: WPAI: CD is a questionnaire used to evaluate lost productivity due to CD ; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Total work productivity impairment takes into account both hours missed due to CD symptoms and the patient's assessment of the degree to which CD affected their productivity while working (overall work impairment [OWI]). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: From first dose of Humira up to 3 years
Population: Efficacy Analysis Set: patients who have assessments at the first administration and the subsequent assessment
Measure: Mean (Standard Deviation); unit: Percent overall work impairment
Arm/Group | Humira
Number analyzed (Participants) | 310
Percent overall work impairment
  At first administration: number analyzed (Participants) | 102
  At first administration | 42.68 (34.71)
  Week 4 of administration: number analyzed (Participants) | 84
  Week 4 of administration | 26.89 (28.45)
  Month 3 of administration: number analyzed (Participants) | 73
  Month 3 of administration | 25.85 (30.40)
  Month 6 of administration: number analyzed (Participants) | 60
  Month 6 of administration | 20.17 (28.63)
  Year 1 of administration: number analyzed (Participants) | 55
  Year 1 of administration | 23.89 (30.43)
  Year 1 and Month 6 of administration: number analyzed (Participants) | 36
  Year 1 and Month 6 of administration | 27.64 (33.18)
  Year 2 of administration: number analyzed (Participants) | 24
  Year 2 of administration | 22.83 (26.22)
  Year 2 and Month 6 of administration: number analyzed (Participants) | 22
  Year 2 and Month 6 of administration | 19.77 (29.93)
  Year 3 of administration: number analyzed (Participants) | 17
  Year 3 of administration | 14.27 (25.06)

6. Secondary Outcome: Change in WPAI: CD Activity Impairment Over Time
Description: WPAI: CD is a questionnaire used to evaluate lost productivity due to CD ; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Activity impairment (percentage of activity impairment due to CD ) is calculated as the patient's rating of how much CD affected their ability to do regular daily activities, other than working at a job (0 = no effect; 10 = completely prevented from working) / 10 * 100. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: From first dose of Humira up to 3 years
Population: Efficacy Analysis Set: patients who have assessments at the first administration and the subsequent assessment
Measure: Mean (Standard Deviation); unit: Percent activity impairment
Arm/Group | Humira
Number analyzed (Participants) | 310
Percent activity impairment
  At first administration: number analyzed (Participants) | 185
  At first administration | 50.22 (31.45)
  Week 4 of administration: number analyzed (Participants) | 167
  Week 4 of administration | 29.22 (26.64)
  Month 3 of administration: number analyzed (Participants) | 130
  Month 3 of administration | 26.46 (26.82)
  Month 6 of administration: number analyzed (Participants) | 112
  Month 6 of administration | 23.66 (25.22)
  Year 1 of administration: number analyzed (Participants) | 85
  Year 1 of administration | 21.76 (24.36)
  Year 1 and Month 6 of administration: number analyzed (Participants) | 63
  Year 1 and Month 6 of administration | 26.51 (25.98)
  Year 2 of administration: number analyzed (Participants) | 46
  Year 2 of administration | 21.52 (21.91)
  Year 2 and Month 6 of administration: number analyzed (Participants) | 43
  Year 2 and Month 6 of administration | 24.88 (25.01)
  Year 3 of administration: number analyzed (Participants) | 26
  Year 3 of administration | 14.62 (18.60)

7. Secondary Outcome: Percentage of Participants With Endoscopic Remission Over Time by Intestine Segment (Large Intestine, Small Intestine, and Both Large and Small Intestine)
Description: Endoscopic remission per endoscopy sub score.
Time Frame: From first dose of Humira up to 3 years
Population: Efficacy Analysis Set: patients who have assessments at the first administration and the subsequent assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Humira
Number analyzed (Participants) | 310
Participants
  Large intestine: start of administration: number analyzed (Participants) | 129
  Large intestine: start of administration | 20
  Large intestine: Month 6 of administration: number analyzed (Participants) | 39
  Large intestine: Month 6 of administration | 17
  Large intestine: Year 1 of administration: number analyzed (Participants) | 64
  Large intestine: Year 1 of administration | 31
  Large intsetine: Year 2 of administration: number analyzed (Participants) | 61
  Large intsetine: Year 2 of administration | 35
  Large intestine: Year 3 of administration: number analyzed (Participants) | 56
  Large intestine: Year 3 of administration | 36
  Small intestine: at first administration: number analyzed (Participants) | 97
  Small intestine: at first administration | 7
  Small intestine: Month 6 of administration: number analyzed (Participants) | 28
  Small intestine: Month 6 of administration | 15
  Small intestine: Year 1 of administration: number analyzed (Participants) | 52
  Small intestine: Year 1 of administration | 25
  Small intestine: Year 2 of administration: number analyzed (Participants) | 46
  Small intestine: Year 2 of administration | 16
  Small intestine: Year 3 of administration: number analyzed (Participants) | 41
  Small intestine: Year 3 of administration | 19
  Both intestine: start of administration: number analyzed (Participants) | 73
  Both intestine: start of administration | 2
  Both intestine: Mont 6 of administration: number analyzed (Participants) | 18
  Both intestine: Mont 6 of administration | 5
  Both intestine: Year 1 of administration: number analyzed (Participants) | 41
  Both intestine: Year 1 of administration | 16
  Both intestine: Year 2 of administration: number analyzed (Participants) | 32
  Both intestine: Year 2 of administration | 8
  Both intestine: Year 3 of administration: number analyzed (Participants) | 26
  Both intestine: Year 3 of administration | 11

8. Secondary Outcome: Change in C-Reactive Protein (CRP) Levels Over Time
Description: CRP values were measured as an inflammatory parameter. Low CRP values mean less inflammation.
Time Frame: From first dose of Humira up to 3 years
Population: Efficacy Analysis Set: patients who have assessments at the first administration and the subsequent assessment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Humira
Number analyzed (Participants) | 310
mg/dL
  At first administration: number analyzed (Participants) | 293
  At first administration | 1.53 (2.00)
  Week 4 of administration: number analyzed (Participants) | 260
  Week 4 of administration | 0.43 (0.99)
  Month 3 of administration: number analyzed (Participants) | 216
  Month 3 of administration | 0.55 (1.09)
  Month 6 of administration: number analyzed (Participants) | 194
  Month 6 of administration | 0.53 (1.18)
  Year 1 of administration: number analyzed (Participants) | 214
  Year 1 of administration | 0.54 (1.00)
  Year 1 and Month 6 of administration: number analyzed (Participants) | 193
  Year 1 and Month 6 of administration | 0.49 (1.31)
  Year 2 of administration: number analyzed (Participants) | 153
  Year 2 of administration | 0.44 (1.03)
  Year 2 and Month 6 of administration: number analyzed (Participants) | 151
  Year 2 and Month 6 of administration | 0.52 (1.38)
  Year 3 of administration: number analyzed (Participants) | 145
  Year 3 of administration | 0.66 (2.90)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from the first dose of study drug until the end of the study (up to 160 weeks).
Description: TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Humira
All-Cause Mortality (participants affected / at risk) | 3/389
Serious Adverse Events (participants affected / at risk) | 58/389
Other Adverse Events (participants affected / at risk) | 104/389
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humira (N=389)
Endocarditis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2)
Respiratory tract infection fungal (Infections and infestations) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Tetany (Metabolism and nutrition disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 8 (8)
Ileal stenosis (Gastrointestinal disorders) | 4 (4)
Ileus (Gastrointestinal disorders) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Intestinal stenosis (Gastrointestinal disorders) | 4 (4)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Subileus (Gastrointestinal disorders) | 1 (1)
Small intestinal stenosis (Gastrointestinal disorders) | 4 (4)
Fistula of small intestine (Gastrointestinal disorders) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Collagen disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1)
Haemorrhoid operation (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humira (N=389)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (8)
Peritonitis (Infections and infestations) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2)
Postoperative wound infection (Infections and infestations) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tracheobronchitis mycoplasmal (Infections and infestations) | 1 (1)
Urethritis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 3 (3)
Psoas abscess (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 2 (2)
Respiratory tract infection fungal (Infections and infestations) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4)
Seasonal allergy (Immune system disorders) | 1 (1)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Tetany (Metabolism and nutrition disorders) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Aortitis (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 8 (8)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 1 (1)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3)
Jaundice (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Collagen disorder (Musculoskeletal and connective tissue disorders) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 2 (2)
Injection site reaction (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Injection site swelling (General disorders) | 3 (3)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 12 (12)
Chest X-ray abnormal (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2)
Blood beta-D-glucan increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Pancreatic enzymes increased (Investigations) | 1 (1)
Antinuclear antibody increased (Investigations) | 1 (1)
Double stranded DNA antibody positive (Investigations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT01464333/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT01464333/SAP_001.pdf